CLINICAL TRIAL: NCT03004534
Title: A Presurgical Tissue-Acquisition Study to Evaluate Molecular Alterations in Human Breast Cancer Tissue Following Short-Term Exposure to the Androgen Receptor Antagonist Darolutamide (ODM-201)
Brief Title: A Study to Evaluate Changes in Human Breast Cancer Tissue Following Short-Term Use of Darolutamide
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Translational Research in Oncology (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRIO030; 2016-004151-79 (EudraCT Number); HC6-24-c 201058 (Other: Health Canada)
Record Dates: First submitted 2016-12-21; First posted 2016-12-29 (Estimated); Results first posted 2020-04-03 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-03

CONDITIONS: Breast Cancer Female
Keywords: Breast Cancer; Breast Carcinoma; Breast Tumours; Early Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — darolutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Presurgical Molecular Assessment (Experimental): Oral 300 mg darolutamide tablet; dose of 600 mg (2 x 300 mg tablets) b.i.d.
  Interventions: Drug: darolutamide

INTERVENTIONS:
Drug: darolutamide — Oral 300 mg tablets; 600 mg (2 x 300 mg tablets) taken twice per day, to a daily dose of 1200 mg.
  Other Names: BAY 1841788; ODM-201

SUMMARY:
The purpose of this study is to evaluate the effect of short-term treatment with darolutamide on breast cancer cells (i.e., how the treatment may change the genes or proteins in breast cancer cells) and to evaluate its safety and the way it is tolerated by subjects.

The intent is to study these changes in order to have a better understanding of the potential use of darolutamide for women with EBC, know which patients are likely or unlikely to respond to this treatment, and determine how darolutamide may be combined with other anti-cancer drugs.

DETAILED DESCRIPTION:
This current study will enroll EBC subjects with differing breast cancer (BC) subtypes, with the intent of characterizing the molecular alterations in BC tissue before and after short-term exposure to the anti-androgen darolutamide. Studying the biological mechanisms in which darolutamide targets the androgen receptor (AR) in BC will be crucial in understanding its' potential role, as well as provide the foundation for further development of darolutamide in this disease.

TRIO030 will evaluate the following objectives: Primary -To identify the molecular alterations that occur in human BC tissue, following short-term exposure to darolutamide in female subjects with EBC; Secondary - To evaluate the safety and tolerability of short-term exposure to darolutamide in female subjects with EBC.

Design: This will be a multi-center, open-label, tissue-acquisition study involving up to 60 subjects from approximately 20 sites in North America and Europe, and will enroll EBC subjects of differing subtypes (i.e., triple negative [TNBC], ER+/HER2-, and HER2+), with the intent of characterizing the molecular alterations in BC tissue before and after short-term exposure to the anti-androgen darolutamide.

Such information may suggest that darolutamide be combined with other modalities; for example, if treatment with the drug is discovered to affect multiple signaling pathways. Molecular profiling of tumor samples before and after darolutamide treatment may permit the identification of patients likely or unlikely to respond to the agent based on the biological and molecular characteristics of their tumors.

Duration: It is recommended that the surgery date is defined prior to starting protocol treatment and then the start date of darolutamide (Day 1) will be derived as minus 14 to 21 days from the scheduled surgery date. Treatment will be taken until the day prior to surgery or when the subject is ordered to stop all oral intake (i.e., "nil per os" (npo)), which ever occurs first. If for some reason surgery takes place more than 21 days after treatment start, it is acceptable that the subject receives darolutamide for more than 21 days and up to a maximum of 35 days; subject should continue protocol treatment until the day prior to surgery, or npo is ordered. In these cases it is strongly recommended to have surgery performed as soon as possible after 21 days of treatment are completed.

After surgery, an End of Study (EoS) visit will occur 30 days (+/- 3 days) after the subject's last intake of darolutamide. In case of ongoing protocol treatment-related AEs/SAEs at the time of the EoS visit, monitoring of these events will continue as clinically indicated until (a) the events have resolved or (b) the events have reached a status which, in the Investigator's opinion, is unlikely to resolve due to the nature of the condition and/or the subject's underlying disease.

Total Number of Sites: A total of 14 sites were opened worldwide, with 5 sites located within the U.S, 6 in Canada, and 3 in Germany.

Sample Size/Patient Population: Up to 60 subjects will be enrolled in the study. To be able to assess the molecular alterations after darolutamide, exposure in different BC subtypes, subjects being either triple-negative, or ER+/HER2 negative, or HER2 positive, will be enrolled in the study. Up to 20 subjects with each of these subtypes will be included (with an acceptable minimum of 8 evaluable patients in each cohort).

Dosage Regimen: Darolutamide will be given at a dose of 600 mg (2 x 300 mg tablets) twice daily (b.i.d) to a daily dose of 1200 mg.

The first day of darolutamide administration in the study is considered Day 1. The last darolutamide intake will be on the day prior to breast cancer surgery, when the pre-surgery visit should occur.

darolutamide should be taken approximately at the same time each day twice a day. It is recommended that darolutamide be taken with food; recommendation is to take it with breakfast and dinner each day.

Supportive measures and dose modifications: A subject who experiences a treatment-related grade 3 or higher adverse event (AE) must be withdrawn from protocol treatment and should proceed to surgery and undergo an EoS visit. In the case of a grade 1-2 treatment-related AE, the Investigator should contact the Medical Monitor if a dose reduction or treatment hold is required.

Washout pre-trial: Prior treatment of ovarian hormone replacement therapy should be stopped at least 28 days prior to registration. Use of other investigational drugs should be stopped within 28 days of enrollment. No major surgery within 28 days before enrollment (Major surgery is defined as requiring a general anesthesia or respiratory assistance; involving openings into the great cavities of the body, organs removed, or normal anatomy altered; implying risks of severe hemorrhage; implying risk for life of the patient or severe disability).

Concomitant Medication: Subjects will be instructed to consult with the Investigator before taking any medications (including over-the-counter medications). Supportive medications may be provided prophylactically or therapeutically per Investigator discretion.

Any concomitant treatment NOT listed below is considered permitted in the study and may be prescribed as clinically appropriate during the study:

* Investigational agents other than the protocol treatment.
* Any additional standard or investigational anticancer agents, such as chemotherapy, immunotherapy, targeted/biologic therapy, endocrine therapy, etc., even if utilized as treatment of non-cancer indications. darolutamide must be permanently discontinued upon initiation of a non-protocol standard or investigational antineoplastic therapy prior to surgery.

Rescue Medication and Risk Management: No specific pre-medication is required. Based on the current available data , there are no special warnings and precautions associated with the use of darolutamide.

Premature Withdrawal / Discontinuation Criteria: The patient may withdraw from the study at any time without prejudicing future medical treatment. In any case, the withdrawal should be clearly documented in the subject's clinical records.

Should a patient decide to withdraw consent, all efforts will be made to complete and report the observations as thoroughly as possible. A complete final evaluation at the time of the patient's withdrawal should be made with an explanation of why the patient is withdrawing from the study. After complete withdrawal of consent, no further study procedure is performed and no further data will be collected.

Discontinuation: The Investigator will also discontinue protocol treatment if any of the following conditions is met:

* Intercurrent illness or a change in subject´s condition or unacceptable toxicity that warrants protocol treatment discontinuation according to Investigator's judgment
* Any event, condition, criterion which would warrant discontinuation of darolutamide (i.e., severe toxicities), including grade ≥ 3 protocol-treatment related AE
* Any event, condition, reason which would warrant darolutamide to be held for more than the maximum acceptable delay of 7 consecutive days
* Subject receives non-protocol anti-cancer therapy at any time during the protocol treatment
* Subject's decision to withdraw protocol treatment
* Lost to follow up
* Death
* Pregnancy
* Investigator's decision
* Discontinuation of the study by the sponsor
* Patient is enrolled but does not receive protocol treatment for any reason

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated PICF obtained prior to initiation of any study-specific procedure and treatment.
2. Female ≥ 18 years old.
3. Histologically proven invasive breast carcinoma (through either a core needle biopsy or an incisional biopsy) for which surgery is indicated as the primary treatment modality. Patients for which Neoadjuvant Systemic Therapy (NAST) is indicated are also eligible provided they are willing to undergo a biopsy after completing treatment with darolutamide and prior to NAST start.
4. Known ER, PgR and HER2 statuses.
5. Tumor must be confined to either the breast or to the breast and ipsilateral axilla (Note: patinets with multifocal/multicentric tumors are eligible). Patient must have (according to TNM 7th edition rules):

   * T1 with T ≥1.0cm, T2 or T3 by at least one radiographic or clinical measurement
   * Either clinically positive (N1 only) or clinically negative axillary nodes (N0)
   * M0
6. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1.
7. Adequate organ function within 28 days prior to enrollment, as defined by the following criteria:

   * Hematology: Hemoglobin ≥ 9.0 g/dl; ANC ≥ 1.5 × 109/L; Platelet count ≥ 100 × 109/L
   * Liver function: ALT and AST ≤ 2.5 × ULN; Total bilirubin ≤ 1.5 × ULN (or ≤ 3 times ULN for patients with documented Gilbert's syndrome or for whom indirect bilirubin concentrations suggest an extra-hepatic source of elevation)
   * Renal function: Creatinine ≤ 2.0 × ULN
8. No more than 42 days should elapse from the day study-specific tumor sample is taken at initial diagnosis (or subsequent procedure) to the day of the first intake of darolutamide.
9. Women of childbearing potential (WoCBP)* must agree to use acceptable non-hormonal contraceptive methods of birth control from the day of the screening pregnancy test and up to 3 months after the last intake of darolutamide.
10. For WoCBP* negative serum pregnancy test within 7 days of enrollment.
11. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and biopsies as detailed in the protocol.

    * Note: WoCBP are any women between menarche and menopause who have not been permanently sterilized, capable of procreation. Permanent sterilization includes hysterectomy and/or bilateral oophorectomy and/or bilateral salpingectomy but excludes bilateral tubal ligation/occlusion. Postmenopause is defined as: Bilateral oophorectomy; Age ≥ 60; Age < 60 and amenorrheic for ≥ 12 months in the absence of an alternative medical cause and FSH and estradiol in postmenopausal ranges.

Exclusion Criteria:

1. Any T0, Tis, T1 < 1.0 cm, T4; or N2-3; or M1 BC.
2. Bilateral invasive BC.
3. Patient that underwent excisional biopsy of the primary tumor.
4. Medical indication or patient desire to undergo BC surgery or start NAST prior to completing at least 14 days of treatment with darolutamide, and or refusal of patient to undergo corresponding biopsy in case NAST is planned.
5. Prior or concurrent systemic anticancer therapy for BC treatment(immunotherapy, hormonotherapy, biologic/targeted therapy, chemotherapy, investigational agents).
6. Prior or concurrent ipsilateral radiation therapy for invasive or noninvasive BC.
7. Prior or concurrent treatment or preventative use of any hormonal agent such as aromatase inhibitors (AI), fulvestrant, raloxifene, tamoxifen or other SERM, or with any other hormonal agent used for the treatment or prevention of BC or for any other indication (e.g. osteoporosis).
8. Concurrent use of ovarian hormone replacement therapy. Prior treatment should be stopped at least 28 days prior to registration.
9. Prior or concurrent treatment with AR antagonists or CYP17 enzyme inhibitor.
10. Use of other investigational drug within 28 days of enrollment.
11. Major surgery* within 28 days before enrollment.
12. Any concurrent or previous malignancy within 5 years prior to enrollment except for basal or squamous skin cancer, or carcinoma in situ of the cervix, or other non-invasive/in-situ neoplasm, all of which must have been adequately and radically treated. A patient with previous history of invasive malignancy (other than adequately and radically treated basal or squamous skin cancer) is eligible provided that she has been disease free for more than 5 years.
13. Severe or uncontrolled concurrent disease, infection or comorbidity.
14. Known active viral hepatitis, HIV or chronic liver disease.
15. Other serious illness or medical condition within 6 months before enrollment, including any of the following: Concurrent congestive heart failure NYHA Class III or IV, severe/unstable angina pectoris, myocardial infarction, uncontrolled hypertension, coronary/peripheral artery bypass graft, high-risk uncontrolled arrhythmias, stroke.
16. Any contraindication to oral agents or gastrointestinal disorder or procedure which expects to interfere significantly with absorption of protocol treatment.
17. History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the patient's participation for the full duration of the trial, or is not in the best interest of the patient to participate, in the opinion of the treating investigator.
18. Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
19. Known allergy to darolutamide or any of the excipients.
20. Pregnant or lactating darolutamide. * Note: Major surgery defined as requiring a general anesthesia or respiratory assistance; involving openings into the great cavities of the body, organs removed, or normal anatomy altered; implying risks of severe hemorrhage; implying risk for life of the patient or severe disability.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2019-02-14 (Actual); Study Completion 2019-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Fresco, MD, Study Director — Translational Research in Oncology
Locations (14):
- United States (5):
  - UCLA, Los Angeles, California
  - Valley Breast Care and Women's Health Center, Los Angeles, California
  - Torrance Memorial Physician Network, Cancer Care Associates, Redondo Beach, California
  - Central Coast Medical Oncology, Santa Maria, California
  - UF Health Cancer Center - Orlando Health, Orlando, Florida
- Canada (6):
  - Cross Cancer Institute, Edmonton, Alberta
  - (CIUSSS) de l'Est-de-l'Île-de-Montréal - l'Hôpital Maisonneuve-Rosemont, Montreal, Quebec
  - Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - McGill University Hospital, Montreal, Quebec
  - Centre Hospitalier Affilie Universitaire De Quebec - Hospital Du Saint-Sacrement, Québec, Quebec
- Germany (3):
  - Universitatsklinikum Erlangen, Erlangen
  - Interdisziplinares Onkologisches Zentrum, München
  - Department of Women's Health, Tübingen

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The screening period starts with registration (which is informed consent signature) and ends when the patient is enrolled (following eligibility central review confirmation by TRIO) or screen failed.
Period: Overall Study
Arm/Group | Presurgical Molecular Assessment
Started | 36
Completed | 36
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 36 patients were enrolled in total. The evaluable population was used for the performance of molecular assays - 35 patients were evaluable based on the clinical criteria (of these 34 were evaluable for molecular analysis based on the adequacy of the tumor tissue collected).
Arm/Group | Presurgical Molecular Assessment
Number analyzed (Participants) | 36
Age, Continuous [Median (Full Range); unit: years] | 61.5 [32.0 to 82.0]
Age, Customized [Count of Participants; unit: Participants]
  Adults (18-64 years) | 20
  Adults (65-84 years) | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 31
  Other | 5
Region of Enrollment [Number; unit: participants]
  Canada | 8
  United States | 21
  Germany | 7
Menopausal Status [Count of Participants; unit: Participants]
  Postmenopausal | 27
  Premenopausal | 9
Breast Cancer Sub-Type [Count of Participants; unit: Participants]
  Triple-negative | 7
  HR+/HER2 negative | 20
  HER2 positive | 9
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — The ECOG Scale of Performance Status is a measurement used to describe a patient's level of functioning in terms of their ability to care for themself, daily activity, and physical ability (walking, working, etc.).
  Patients with ECOG 0 are in better general condition than patients with ECOG 1:
  0 = Fully active, able to carry on all pre-disease performance without restriction.
  1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work.
  Participants
    ECOG 0 | 35
    ECOG 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Identifying Molecular Alterations in Breast Cancer Tissue Tumor Samples Following Short-Term Preoperative Exposure to Darolutamide in Female Patients Wit Early Breast Cancer.
Description: Androgen Receptor (AR) was assessed on the collected samples.
Time Frame: 1 year, 6 months
Population: 36 patients were enrolled, however 34 patients were evaluable based on the molecular criteria: Adequacy (evaluated by the central laboratory) for molecular assessment of the tumor tissue collected before and after the protocol treatment initiation. Expression levels were evaluated by microarray using the patient's RNA.
Measure: Count of Participants; unit: Participants
Arm/Group | Presurgical Molecular Assessment
Number analyzed (Participants) | 34
Participants
  Androgen Receptor - Up | 7
  Androgen Receptor - Unchanged | 12
  Androgen Receptor - Down | 15

2. Secondary Outcome: Number of Participants With Treatment-related Adverse Events (TEAE) as Assessed by CTCAE v4.03
Description: The assessment of safety will be performed for all subjects who have taken at least one tablet of darolutamide (defined as the "safety population")
Time Frame: 1 year, 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Presurgical Molecular Assessment
Number analyzed (Participants) | 36
Participants
  No. of Patients with a TEAE | 26
  No. of Patients without a TEAE | 10

ADVERSE EVENTS:
Time Frame: 1 year, 6 months.
Description: The Safety population includes all patients who have taken at least one tablet of darolutamide. The following information was collected: description of event, start/stop dates, worst grade experienced (severity/intensity), seriousness, action taken on protocol treatment, and relationship to protocol treatment. The intensity of AEs were classified and recorded according to NCI CTCAE version 4.03. All adverse experiences observed by the Investigator or reported by the patient were collected.
Arm/Group | Presurgical Molecular Assessment
All-Cause Mortality (participants affected / at risk) | 0/36
Serious Adverse Events (participants affected / at risk) | 0/36
Other Adverse Events (participants affected / at risk) | 26/36
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Presurgical Molecular Assessment (N=36)
Constipation (Gastrointestinal disorders) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 3 (3)
Nasea (Gastrointestinal disorders) | 3 (3)
Fatigue (General disorders) | 8 (8)
Nasopharyngitis (Infections and infestations) | 2 (2)
Upper Respiratory Tract Infection (Infections and infestations) | 2 (2)
Procedural Pain (Injury, poisoning and procedural complications) | 2 (2)
ALAT Increase (Investigations) | 2 (2)
ASAT Increase (Investigations) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Dysuria (Renal and urinary disorders) | 2 (2)
Breast Pain (Reproductive system and breast disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication, abstract or presentation of the study will be made without the approval of the Study Steering Committee (SSC).

DOCUMENTS (2):
  • Study Protocol (2018-02-16): https://cdn.clinicaltrials.gov/large-docs/34/NCT03004534/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-30): https://cdn.clinicaltrials.gov/large-docs/34/NCT03004534/SAP_001.pdf